CLINICAL TRIAL: NCT00393003
Title: Target-controlled Infusion of Propofol and Remifentanil for Postoperative Sedation Guided by the Bispectral Index: Comparison Between Manual Perfusion and Automated Perfusion
Brief Title: Target-controlled Infusion of Propofol and Remifentanil for Postoperative Sedation Guided by the Bispectral Index
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Marc Fischler, Hopital Foch
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Foch-1
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2009-08-31 (Estimated); Status verified 2009-08

CONDITIONS: Postoperative Sedation
Keywords: Anesthesia; Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Closed-loop anesthesia system

SUMMARY:
This prospective randomized study evaluates the effectiveness of a closed-loop anesthesia system during the postoperative period.

DETAILED DESCRIPTION:
The Bispectral Index (BIS) is an electroencephalogram-derived measure of anesthetic depth. A closed-loop anesthesia system can be built using BIS as the control variable, two proportional-integral-differential control algorithms, a propofol and a remifentanil target-controlled infusion systems as the control actuators. Preliminary results show that this system can be used during surgery. We propose a prospective randomized study to evaluate the effectiveness of such a closed-loop anesthesia system during the postoperative period. Two groups of patients are compared: one in which propofol and remifentanil are administered by the anesthesiologist using target-controlled infusion systems, and one in which propofol and remifentanil are administered automatically by the combined closed-loop anesthesia system. In both groups, the goal is to maintain BIS between 40 and 60, the recommended range during anesthesia by the manufacturer. We expect the combined closed-loop system group to do similar or better.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1-3
* Abdominal aorta surgery

Exclusion Criteria:

* Pregnant women
* Neurological or muscular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Global score (calculated parameter which depicts the performance of the system)

SECONDARY OUTCOMES:
Consumption of propofol and remifentanil, modifications of target of propofol and remifentanil, dysfunction of each system, hemodynamic abnormalities, sedation scale, volume loading, extubation time, explicit memorisation.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Dept of Anesthesia and Intensive Care, Hopital Pitié-Salpêtrière, 75013 Paris, France
Locations (2):
- France (2):
  - Dept of Anesthesia and Intensive Care, Hopital Pitié-Salpêtrière, Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963